CLINICAL TRIAL: NCT01950195
Title: A Pilot Study of Stereotactic Radiosurgery Combined With Ipilimumab in Patients With Newly Diagnosed Melanoma Metastases in the Brain and Spine
Brief Title: SRS (Stereotactic Radiosurgery) Plus Ipilimumab
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Local IRB required us to submit amendment as a separate study.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1382
Record Dates: First submitted 2013-06-21; First posted 2013-09-25 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Newly Diagnosed Melanoma Metastases in the Brain and Spine
Keywords: Melanoma; Metastases; Brain; Spine; SRS(Stereotactic Radiosurgery)); Ipilimumab
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — Radiosurgery; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brain (Experimental): A cohort of six (6) patients will be treated at Dosing Schedule 1. If the observed dose limiting toxicity (DLT) rate is less ≤33%, the dose cohort will be expended to a total of 15 patients. Brain and spine metastases will be evaluated as two separate cohorts.
  If the first schedule produces DLTs in >33% of patients, the Second Dosing schedule will be implemented. If the second dosing schedule produces DLTs in >33% of patients, the Third Dosing schedule will be implemented.
  After 6 patients were enrolled in a cohort, their safety and toxicity will be continuously monitored till 12 weeks (3 months) after the initial dose of Ipilimumab is given for evaluating dose-limiting toxicities.
  Interventions: Procedure: Stereotactic Radiosurgery (SRS); Biological: Ipilimumab
- Spine (Experimental): A cohort of six (6) patients will be treated at Dosing Schedule 1. If the observed dose limiting toxicity (DLT) rate is less ≤33%, the dose cohort will be expended to a total of 15 patients. Brain and spine metastases will be evaluated as two separate cohorts.
  If the first schedule produces DLTs in >33% of patients, the Second Dosing schedule will be implemented. If the second dosing schedule produces DLTs in >33% of patients, the Third Dosing schedule will be implemented.
  After 6 patients were enrolled in a cohort, their safety and toxicity will be continuously monitored till 12 weeks (3 months) after the initial dose of Ipilimumab is given for evaluating dose-limiting toxicities.
  Interventions: Procedure: Stereotactic Radiosurgery (SRS); Biological: Ipilimumab

INTERVENTIONS:
Procedure: Stereotactic Radiosurgery (SRS)
Biological: Ipilimumab

SUMMARY:
This research is being done to look at the safety of using stereotactic radiosurgery (SRS) and Ipilimumab together to treat melanoma that has spread to the brain or spine. Both Ipilimumab and SRS are used alone for the treatment of melanoma that has spread. Standard of care uses both of these treatments but not together. By using them together, we expect better treatment of melanoma, but there might be an increase in side effects.

"Ipilimumab" is approved by the Food and Drug Administration (FDA) for the treatment of melanoma that has spread throughout the body. It works by activating your immune system to fight off cancer.

"Stereotactic radiosurgery" (SRS) is approved by the Food and Drug Administration (FDA) for the treatment of melanoma in the brain or spine. It uses radiation to treat tumors without needing to cut or use stitches.

The use of combining SRS and Ipilimumab in this research study is investigational. The word "investigational" means that this combination is not approved for marketing by the Food and Drug Administration but is allowed for use in this research study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed diagnosis of melanoma. The pathologic confirmation may be from another metastatic site or from metastatic brain or spine lesions.
2. Patients must have Stage IV melanoma, with newly identified brain or spine metastases.
3. Patients must have measurable lesion in the brain or spine that is > 3 mm seen on magnetic resonance imaging (MRI) with contrast.

   NOTE: Contrasted pre-treatment MRI scan must be obtained ≤ 21 days prior to stereotactic radiosurgery treatment.
4. Karnofsky Performance Scale >70%
5. Patients must have normal organ and marrow function as defined below:

   leukocytes >3,000/mcL absolute neutrophil count >1,500/mcL platelets >100,000/mcL total bilirubin ≤2X institutional upper limit of normal AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal creatinine within normal institutional limits OR According to Johns Hopkins MRI policy
6. Women of child bearing potential (WOCBP) using a reliable form of contraception during the study treatment period and for up to 12 weeks following the last dose of study drug [21].
7. Men must agree to the use of male contraception during the study treatment period and for at least 12 weeks after the last dose of study drug.
8. Ability to understand and the willingness to sign written informed consent document(s).

Exclusion Criteria:

1. Prior whole brain radiation or conventional radiation to the spine at the site of new lesion.
2. Prior chemotherapy within 28 days of starting treatment.
3. Prior therapy with investigational drugs within 28 days or at least 5 half-lives (whichever is longer) before study administration.
4. Prior therapy with an anti-PD-1, anti-PD-L1, anti-PDL-2, or anti-CTLA-4 antibody.
5. Neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
6. Known allergy to compounds of similar chemical or biologic composition to ipilimumab.
7. Pregnant or breastfeeding women.
8. Known history of Human Immunodeficiency Virus.
9. Active infection requiring therapy, positive tests for Hepatitis B surface antigen or Hepatitis C ribonucleic acid (RNA) [11].
10. Active autoimmune disease, history of autoimmune disease or history of syndrome that required systemic steroids or immunosuppressive medications. Exceptions include those with vitiligo or resolved childhood asthma/atopy. Subjects with asthma who require intermittent use of bronchodilators (such as albuterol) will not be excluded from this study [11].
11. Use of any vaccines against infectious diseases (e.g. varicella, influenza, etc.) up to 4 weeks (28 days) before receiving ipilimumab.
12. Prisoners or subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness.
13. Patients with both brain and spine metastases will be excluded from the trial.
14. Patients who are allergic to MRI contrast agent or have contraindication for MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-09; Primary Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of adverse events and severity of the adverse events. | 2 years
  To assess the safety profile of stereotactic radiosurgery with ipilimumab in combination to treat patients with newly diagnosed melanoma brain or spinal metastases.

SECONDARY OUTCOMES:
To estimate local control rate in brain and spine | 1 years
  To estimate systematic control rate; To estimate progression-free survival

OTHER OUTCOMES:
Correlative Objective | 3 years
  To explore peripheral blood immune response during and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lim, MD, Principal Investigator — Johns Hopkins Department of Neurosurgery
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States